CLINICAL TRIAL: NCT00683683
Title: The Strategies for Post Arrest Resuscitation and Care Network
Acronym: SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Laerdal Medical (Industry)
Responsible Party: Principal Investigator, Laurie Morrison, Director, Rescu, Unity Health Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARC (Morrison 038-2008)
Record Dates: First submitted 2008-05-15; First posted 2008-05-23 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-05

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest, hypothermia, knowledge translation
MeSH Terms: conditions — Heart Arrest; Hypothermia | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cooling (Other): Cardiac arrest patients will be cooled to 32-34°C within 6 hours of ED arrival
  Interventions: Behavioral: Knowledge Translation

INTERVENTIONS:
Behavioral: Knowledge Translation — The multifaceted KT strategy will include 1) local multidisciplinary champions in ED, ICU, and Cardiology 2) A simple protocol for application of hypothermia, tailored to local needs and policy; 3) Identification of perceived and actual barriers to knowledge use; 4) Development of an implementation tool kit and 5) Providing timely feedback on benchmarks for hypothermia and outcomes.
  Other Names: Clinical Protocol;; Reminders;; Audit & Feedback;; Network

SUMMARY:
Background: One of the 2010 Impact Goals of the Emergency Cardiac Care (ECC) Committee of the American Heart Association is to double survival from cardiac arrest. Currently, approximately 60% of adults and 50% of paediatric patients that regain spontaneous circulation following cardiac arrest die before leaving the hospital. A key piece of the "chain of survival" is this fifth link; the care of patients post-arrest. Although there are several modalities recommended for post arrest care, therapeutic hypothermia is the only in-hospital therapy that has been demonstrated in randomized clinical trials to improve patient outcome after cardiac arrest. Despite the strong evidence for its efficacy and the apparent simplicity of this intervention, recent surveys show that hypothermia is delivered inconsistently, incompletely, and with undue delay in hospitals receiving resuscitated patients; only 26% of physicians and 26% of hospitals regularly institute a hypothermia protocol.

Primary Objective: To design and apply a knowledge translation program for the 2005 AHA guideline on hypothermia post cardiac arrest and enable effective implementation of hypothermia in 100% of eligible OHCA patients. The integration of two robust data collection systems, which include both pre-hospital and in-hospital indicators, will give complete process of care and clinical outcome information for all cardiac arrest patients.

Primary Endpoint: the proportion of eligible out of hospital cardiac arrest patients cooled to 32-34°C within 6 hours of ED arrival.

Study Design: This project will be implemented through an established research collaborative of 43 hospitals in southern Ontario currently participating in the Toronto site of the Resuscitation Outcomes Consortium. A stepped wedge study design will be employed, whereby the intervention will be rolled-out sequentially to the participating hospitals over a number of time periods as sites reach pre-defined benchmarks. The multifaceted KT strategy will include 1) local multidisciplinary champions in ED, ICU, and Cardiology 2) A simple protocol for application of hypothermia, tailored to local needs and policy; 3) Identification of perceived and actual barriers to knowledge use; 4) Development of an implementation tool kit and 5) Providing timely feedback on benchmarks for hypothermia and outcomes

DETAILED DESCRIPTION:
Substantial resources are spent in providing emergency medical services to victims of out-of-hospital cardiac arrest. The science of pre-hospital medicine has advanced considerably over the past decade. Specifically, EMS services and medical directors have developed carefully designed protocols, intensive training, and very substantial resources, in attempting to improve the immediate outcomes in patients with out-of-hospital cardiac arrest. It is anticipated that approximately 200-400 patients per year in the Greater Toronto Area are successfully resuscitated by Emergency Medical Services personnel and be admitted to hospital with intact circulatory function.

Unfortunately, many of these patients will then die following hospital admission, from one of a variety of complications of the initial cardiac arrest. The "in-hospital attrition rate" is approximately 50%, and is the result of short and longer-term organ damage suffered during the circulatory arrest, as well as in-hospital complications including pulmonary, neurological, septic, and multi-organ dysfunction related complications.

Although guidelines for specific aspects of intensive care therapy of critically ill patients have been developed (for example, ventilation guidelines, sepsis prevention and therapy guidelines, treatment of metabolic disorders, etc), practical guidelines, which are specifically aimed at the investigation and treatment of patients resuscitated from out-of-hospital cardiac arrest, do not currently exist.

Preliminary studies (in press) suggest that a program of comprehensive and consistent adherence to a specific set of standard procedures in intensive care units can lead to a substantial improvement in the survival of patients resuscitated from cardiac arrest. One recent example is a study from Oslo Norway, which showed substantial improvements in survival to discharge following out-of-hospital cardiac arrest after a set of informal guidelines were adopted by participating intensive care units.

There are multiple reasons for the lack of clearly articulated guidelines and protocols for the investigation and treatment of patients resuscitated following cardiac arrest however the two most obvious are lack of understanding of the current recommended best practices and practical impediments to their efficient implementation in all units.

The Resuscitation Outcomes Consortium (ROC), an NIH funded multi-centre effort, seeks to randomize over 10,000 patients in selected North American sites to study specific interventions designed to improve long term survival in patients with out-of-hospital cardiac arrest. As part of this consortium, intensive care units in the ROC hospitals are being invited to join a new best practice initiative entitled "Strategies for Post Arrest Care in the ICU" (SPARC).

Working with more than 50 hospitals across Ontario, the objectives of the SPARC Project are planned as follows:

1. To establish a network of intensive care units, with medical and nursing leaders who will participate in a collaborative program designed to standardize, monitor, and improve the care of patients resuscitated from out-of-hospital cardiac arrest.
2. To develop a series of standardized protocols and processes for the care of patients following out-of-hospital cardiac arrest, with particular emphasis on the delivery of post cardiac arrest mild hypothermia. These protocols will be based on best evidence to date and will focus on the simplifying the processes required implement the recommended interventions.
3. To conduct pragmatic clinical trials of the integrated post cardiac arrest protocol versus historical controls, and study related patient outcomes such as survival to hospital discharge. We will also look to provide a comprehensive assessment of in-hospital complications, the incidence of presumed myocardial ischemic events causing cardiac arrest, and to assess the causes of in-hospital and post discharge morbidity and mortality for the one year following discharge, as a function of the presumed underlying cause of cardiac arrest and the in-hospital course.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals participating in the ROC network

Exclusion Criteria:

* Hospitals who do not receive out-of-hospital cardiac arrest patients

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible out of hospital cardiac arrest patients cooled to 32-34°C within 6 hours of ED arrival. | Within 6 hours of ED arrival.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Morrison, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre

REFERENCES:
- [Derived] Morrison LJ, Brooks SC, Dainty KN, Dorian P, Needham DM, Ferguson ND, Rubenfeld GD, Slutsky AS, Wax RS, Zwarenstein M, Thorpe K, Zhan C, Scales DC; Strategies for Post-Arrest Care Network. Improving use of targeted temperature management after out-of-hospital cardiac arrest: a stepped wedge cluster randomized controlled trial. Crit Care Med. 2015 May;43(5):954-64. doi: 10.1097/CCM.0000000000000864. PMID 25654175
- [Derived] Dainty KN, Scales DC, Brooks SC, Needham DM, Dorian P, Ferguson N, Rubenfeld G, Wax R, Zwarenstein M, Thorpe K, Morrison LJ. A knowledge translation collaborative to improve the use of therapeutic hypothermia in post-cardiac arrest patients: protocol for a stepped wedge randomized trial. Implement Sci. 2011 Jan 14;6:4. doi: 10.1186/1748-5908-6-4. PMID 21235799